CLINICAL TRIAL: NCT07229547
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Safety and Efficacy of Onradivir Tablets in Participants Aged 12 to 17 Years With Uncomplicated Influenza A.
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RuijinH
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): Placebo Group:
  Take the Onradivir Tablets matching placebo once daily, 3 tablets per dose, for a total of 5 days (5 doses).
  Interventions: Drug: Placebo
- Onradivir Tablet Group (Experimental): Onradivir Tablets Group:
  Take Onradivir Tablets once daily, 600 mg (3 tablets) per dose, for a total of 5 days (5 doses).
  Interventions: Drug: Onradivir tablet

INTERVENTIONS:
Drug: Placebo — A placebo that resembles Onradivir tablet in appearance, weight, and odor. The external packaging of Onradivir tablet and the placebo is identical. Take placebo once daily, 3 tablets per dose, for a total of 5 days (5 doses).
  Arms: Placebo Group
Drug: Onradivir tablet — Take Onradivir Tablets once daily, 600 mg (3 tablets) per dose, for a total of 5 days (5 doses).
  Arms: Onradivir Tablet Group

SUMMARY:
This randomized, double-blind, placebo-controlled study is designed to evaluate the efficacy and safety of Onradivir Tablets in participants aged 12 to 17 years with influenza A virus infection.

The trial plans to enroll approximately 150 adolescent participants (12-17 years) with uncomplicated influenza A, confirmed by rapid antigen/nucleic acid testing and within 48 hours of symptom onset. Eligible participants who meet the inclusion criteria and do not meet any exclusion criteria will be randomized in a 2:1 ratio to receive either Onradivir Tablets or placebo once daily for 5 consecutive days.

The study consists of a screening period, a treatment period, and a safety follow-up period. Each participant will be followed up until Day 14 after the first dose. Nasopharyngeal swabs will be collected at screening, Day 2, Day 4, Day 5, and Day 10 for virological testing, including:

Viral load measurement by reverse transcription quantitative polymerase chain reaction (RT-qPCR)

Viral titer determination by culture assay (50% tissue culture infectious dose, TCID₅₀)

Throughout the treatment and safety follow-up periods, participants will record body temperature, influenza symptom scores, and daily activity scores using a diary card. Clinical laboratory tests will be performed at screening, Day 5, and Day 15. Physical examinations and vital signs measurements will be conducted at each follow-up visit. Adverse events and concomitant medications will be documented throughout the study.

ELIGIBILITY:
Inclusion Criteria:

-

All participants must meet all of the following criteria:

Aged 12 to 17 years (inclusive), regardless of gender.

Diagnosed with influenza A based on the following criteria:

* Positive for influenza A virus infection by Rapid Antigen Test (RAT) or nucleic acid testing of nasopharyngeal/oropharyngeal swab at screening.
* Axillary temperature ≥38°C at screening. If this criterion is not met due to antipyretic use, reassessment may be performed >4 hours after the most recent antipyretic administration.
* Presence of at least one moderate or severe influenza-related systemic symptom (headache, fever or chills, muscle or joint pain, fatigue) at screening.
* Presence of at least one moderate or severe influenza-related respiratory symptom (cough, sore throat, nasal congestion) at screening.

Onset of the first influenza symptom/sign occurring within ≤48 hours before randomization. Influenza symptoms/signs include fever (based on participant-reported data, body temperature ≥37.5°C), headache, muscle or joint pain, fatigue, cough, sore throat, and nasal congestion.

Participant's parent/legal guardian and the participant themselves provide signed informed consent before the trial, with full understanding of the trial content, procedures, and potential adverse reactions.

In the investigator's judgment, the participant and their parent/legal guardian are willing and able to comply with the study protocol requirements.

Exclusion Criteria:

* Participants will be excluded from the study if they meet any of the following criteria:

Judged by the investigator as having severe or critical influenza.

Having allergic constitution, known allergy to Anladiwei or paracetamol, and/or clinically suspected intolerance, or having contraindications.

Difficulty swallowing the investigational product, or history of gastrointestinal diseases that severely affect drug absorption (including but not limited to reflux esophagitis, chronic diarrhea, inflammatory bowel disease, intestinal tuberculosis, gastrinoma, short bowel syndrome, partial gastrectomy, etc.).

History of febrile seizures.

High-risk population for severe cases, defined as having any of the following conditions:

* Respiratory diseases judged clinically significant by the investigator (e.g., interstitial lung disease, pulmonary hypertension, cystic fibrosis, asthma), metabolic diseases, hematological diseases, cardiovascular and cerebrovascular diseases, liver diseases, kidney diseases, neurological and neuromuscular diseases, psychiatric disorders, or other serious underlying conditions.
* Immunocompromised status, such as malignant tumors, organ or bone marrow transplantation, HIV infection, or use of systemic immunosuppressants within the past 3 months.

Concurrent conditions requiring treatment with medications containing aspirin or salicylates.

History of allergic diseases requiring regular use of antihistamines or other prohibited medications; or occurrence of acute respiratory infection, bronchitis, otitis media, or sinusitis within 2 weeks before onset (appearance of the first influenza symptom/sign); or presence of respiratory symptoms (cough, nasal congestion, runny nose, sore throat) within 1 week before onset.

Presence of suspected pharyngoconjunctival fever, herpangina, measles, purulent tonsillitis, or other respiratory infectious diseases or communicable diseases.

Suspected co-infection requiring systemic treatment, in addition to influenza A virus infection.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Time to alleviation of influenza symptoms | Up to Day 15

SECONDARY OUTCOMES:
Time to fever resolution | Up to Day 15
  axillary temperature ≤37.2°C
Change from baseline in influenza A viral quantification | Up to Day 15
  Change from baseline in influenza A viral quantification (viral titer and viral RNA load)
Duration of detectable viral titer and viral RNA load | Up to Day 15
Proportion of participants with positive viral titer and viral load | Up to Day 15
Area under the curve of viral quantification versus time | Up to Day 15
  Area under the curve (AUC) of viral quantification (viral titer and viral RNA load) versus time
Incidence of influenza-related complications | Up to Day 15
  Incidence of influenza-related complications (hospitalization, death, sinusitis, bronchitis, otitis media, pneumonia, myocarditis, pericarditis, neurological complications, musculoskeletal complications, etc.)
Proportion of participants with symptom resolution | Up to Day 15
Time to resolution of systemic symptoms | Up to Day 15
  Time to resolution of systemic symptoms (headache, fever or chills, muscle or joint pain, fatigue)
Time to resolution of respiratory symptoms | Up to Day 15
  Time to resolution of respiratory symptoms (cough, sore throat, nasal congestion)
Time to resolution of individual symptoms | Up to Day 15
Proportion of participants with fever resolution | Up to Day 15
Proportion and frequency of participants using symptomatic treatment medications | Up to Day 15
Time to return to normal daily activities | Up to Day 15

IPD SHARING:
Plan to Share IPD: Yes